CLINICAL TRIAL: NCT02129621
Title: Prospective Study of Neutrophil Gelatinase Associated Lipocalin (NGAL)as a Biomarker of Mineralocorticoid Receiver Activity in Human: Proof of Concept.
Brief Title: Search of Biomarkers of Mineralocorticoid Receiver Activity : the Value of Neutrophil Gelatinase Associated Lipocalin (NGAL)in Serum or Urine in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-A01008-45
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Diseases
Keywords: Lipocalin; mineralocorticoid receptor
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Urinary and blood lipococalin levels determination — Blood test on an empty stomach. Urinary taking on arrival in the service
Drug: Spironolactone — For the group 5, at the time of the V0 visit, a treatment by aldactone will be set up (posology: 1 to 2 mg/kg).
  Other Names: ALDACTONE

SUMMARY:
Aldosterone and its target the mineralocorticoid receptor are implied in development of cardiovascular disease such as arterial high blood pressure or cardiac failure. Serum aldosterone level is insufficient to know if the mineralocorticoid receptor is activated or not. The aim of this study is to identify biomarkers of mineralocorticoid receptor activity. The first "candidate biomarker" is Neutrophil gelatinase-associated lipocalin (NGAL) or "lipocalin" which being measured in blood or in the urine. According to scientific knowledge's evolution, others biomarkers could be tested later thanks to the blood or urinary samples taken during study.

DETAILED DESCRIPTION:
This study is broken up into 5 groups:

The first is a pre-analytical study to determinate optimum conditions for lipocalin samples.

The second focuses on intra-individual variations of lipocalin levels in blood and urine.

The third determinate the normal values of lipocalin in blood and urine. Fourthly, we study the role of renal function on serum and urines lipocalin levels.

Fifthly, we study the role of anti-aldosterone treatment on patients who suffer of primary hyperaldosteronism.

ELIGIBILITY:
For the group 1 and 2

Inclusion criteria:

* Men having an age ranging between 18 and 35 years
* Unhurt subject of any acute pathology for more than 7 days
* Consent signed by the subject

Exclusion criteria:

* Subject presenting a known arterial high blood pressure (blood pressure > 140/90 mmHg) or any cardiovascular history
* Subject presenting a known renal insufficiency
* Subject presenting a known anaemia (Hb < 12g/dl)
* Subject presenting a known diabetes
* Subject presenting a cancer diagnosed less than 5 years previously or evolutionary cancer
* Subject presenting a chronic liver disease
* Subject presenting a connectivite: Rhumatoid polyarthritis....
* Crohns disease
* Current tuberculosis
* Any medicinal treatment
* Subject participating in another protocol or in exclusion's period for another protocol
* Absence of social insurance

For group 3

Inclusion criteria:

* Men or women having an age ranging between 18 and 85 years
* Unhurt subject of any acute pathology for more than 7 days
* without any cardiovascular treatment
* Consent signed by the subject

Exclusion criteria:

* Subject presenting a known arterial high blood pressure (blood pressure > 140/90 mmHg or > 160/95 mmHg after 60 years)
* Subject presenting a known renal insufficiency
* Subject presenting a known diabetes
* Woman who is pregnant
* Subject presenting a cancer diagnosed less than 5 years previously or evolutionary cancer
* Subject presenting a chronic liver disease
* Subject presenting a connectivite: Rhumatoid polyarthritis....
* Crohns disease
* Current tuberculosis
* Subject presenting an effort angor or other coronaropathy
* Subject with antecedant of endarterectomy of carotid
* Subject with known abdominal aorta aneurism
* Subject participating in another protocol or in exclusion's period for another protocol
* Absence of social insurance

For group 4

Inclusion criteria:

* Men or women having an age ranging between 18 and 85 years
* Subject with chronique renal insufficiency
* Consent signed by the subject

Exclusion criteria:

* Subject presenting a known diabetes
* Woman who is pregnant
* Subject presenting a cancer diagnosed less than 5 years previously or evolutionary cancer
* Subject presenting a chronic liver disease
* Subject presenting a connectivite: Rhumatoid polyarthritis....
* Crohns disease
* Current tuberculosis
* Subject presenting an effort angor or other coronaropathy
* Subject with antecedant of endarterectomy of carotid
* Subject with known abdominal aorta aneurism
* Subject participating in another protocol or in exclusion's period for another protocol
* Absence of social insurance

For the group 5

Inclusion Criteria:

* Men or women having an age ranging between 30 and 60 years
* Hypertensive subject suffering from primary hyperaldosteronism defined by an aldosteron/renin ratio > 64 pmol/mL in position lying and an aldosteron level > 500pmol lying down (or > 550pmol/L seated or standing) or urinary aldosteron level > 63 nmol/24 hours; for whom
* Subjects having an indication for a monotherapy treatment by ALDACTONE (1 or 2 mg/kg/j)during preoperative period, possibly associated if need be with a calcic inhibitive treatment, central or alphabloquant treatment.
* Subject without other cardiovascular history (myocardic infarction, decompensation of cardiac insufficiency, intellectual vascular accident) and with a normal renal function according to the age,the sex and the blood value of creatinine by the formula MDRD (Flow of renal filtration > 60mL/min/1,73)
* Consent signed by the subject

Exclusion Criteria:

* Subject presenting others forms of high blood pressure (consumption of products or medicines which can facilitate or deteriorate the high blood pressure (alcohol, licorise (of whom the "pastis" without alcohol), anti-inflammatory drugs, corticosteroids, ciclosporin, erythropoiétin, cocain), hyperthyroidy, hypercorticism, chronic renal disease: urinary protein level < 0.3 g/l and clearance of the creatinine > 60ml/min/1.73m2), arterial renal stenosis
* Counter -indication of realization of a test of salt injection
* Current pregnancy
* Subject presenting a cancer diagnosed less than 5 years previously or evolutionary cancer
* Chronic liver disease
* Subject presenting a connectivite: Rheumatoid polyarthritis....
* Crohns disease
* Current tuberculosis
* Absence of social insurance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Lipocalin blood and urinary concentrations | 8 months
  Serum and urinary lipocalin concentrations will be evaluated using comercially available kits (Kits lipocalin-2/NGAL (NCAL20))

CONTACTS AND LOCATIONS:
Overall Officials: Michel AZIZI, Pr, Principal Investigator — Georges Pompidou Hospital, Paris
Locations (3):
- France (3):
  - Brabois Hospital, Nancy
  - Georges Pompidou Hospital, Paris
  - Unit of arterial high blood pressure of the Georges Pompidou Hospital, Paris